CLINICAL TRIAL: NCT02562846
Title: Prediction of ECT Treatment Response in Depression and Early Detection of ECT-related Memory Problems
Brief Title: PRediction Of Treatment Response to ECT in Depression and Cognitive Side effecTs
Acronym: PROTECT
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Linda van Diermen, Dr., Universiteit Antwerpen
Other Study IDs: B300201524466
Record Dates: First submitted 2015-08-26; First posted 2015-09-29 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Depression
Keywords: electroconvulsive therapy; response prediction; cognitive side effects
MeSH Terms: conditions — Depression | interventions — Psychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ECT patients: Depressive patients receiving electroconvulsive therapy.
  Interventions: Other: Psychological testing and biological sample collection

INTERVENTIONS:
Other: Psychological testing and biological sample collection — For this study, there will be psychological tests, blood and hair sample collections, and part of the patients will undergo an MRI.

SUMMARY:
It has been convincingly demonstrated that electroconvulsive therapy (ECT) works better and sooner than antidepressants in the treatment of certain subtypes of depression. Given this effectiveness, it would be unfortunate not to give ECT to patients with good response chances as this could substantially shorten the length of a severe depressive episode. Instead of going through all possible psychopharmacological treatment steps, ECT could be proposed much earlier as a treatment option for those patients who might have good response chances. This would be a great advantage for the severely depressed patient, with a decreased disease-burden and hospitalization duration.

However, up to now, objective and reliable predictive factors for good ECT response have not yet been established. Clinical characteristics such as psychomotor retardation, psychotic features and age have often been used to predict the outcome of ECT, but there is too little evidence to consider these as strong predictive factors.

The current project is designed to allow better prediction of ECT-response. The investgators base their selection of predictors on clinical impression and previous research results. The predictive capacity of psychomotor functioning, psychotic symptoms and several biomarkers will be investigated. With these clinical and biological patient and depression characteristics, the investigators aim to develop a decision making tool that will allow a more accurate indication of ECT.

The investigators also investigate ways to predict whether or not a patient will have a good response when treatment has already started, based on an early improvement of psychomotor functioning.

Another subject of great importance is predicting and preventing side-effects. When patients at risk for lasting cognitive side-effects can be identified early in the treatment course, treatment can be adjusted to prevent persistence of memory problems. Therefore, the second part of the study focuses on identifying people at risk for cognitive side effects early in the treatment course.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to PZ Duffel and eligible for ECT because of major depressive disorder of major depressive episode in bipolar disorder (according to DSM-5 criteria).
* Score on HDRS ≥ 17.
* Have signed an IC form indicating that they understand the purpose of and procedures required for the study and are willing to participate in this study. In case of incapacity, a close relative will be asked to give informed consent.
* Be medically stable on the basis of physical examination and vital signs performed during the pre-ECT screening procedure.

Exclusion Criteria:

* Drug or alcohol dependence as detected in the MINI interview at screening (<6 months before ECT).
* Primary psychotic disorder according to DSM-5 criteria (<6 months before ECT).
* Is currently enrolled in a study with an investigational study drug.
* Has any condition that, in the opinion of the investigator, would compromise the wellbeing of the subject or the study or prevent the subject from meeting or performing study requirements.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators include a severely depressed patient population that has to be evaluated regularly. For that reason, the investigators choose residential patients. They are recruited at the psychiatric hospital in Duffel.
  Treating psychiatrists consider a candidate eligible for ECT and start pre-ECT investigations. The investigators screen all depressive ECT patients for inclusion in the study and ask for their informed consent (IC). The treating psychiatrist decides when ECT is stopped considering clinical evolution and side effects.
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2015-06; Primary Completion 2017-09-30 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Change in depression severity as measured by the Hamilton Depression Rating Scale (HDRS) | Baseline measurement before the first electroshock, compared with final HDRS score measured after the last electroshock of the acute ECT course. The duration between the measurement before and after ECT will be between 3-9 weeks.
  The HDRS is one of the most commonly used instruments for assessing depression. It is a valid and reliable clinician-rated measure that has been used extensively in clinical research and in clinical practice for assessment of the severity of depression, changes in its severity over time and efficacy of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Sabbe, MD, prof., Study Director — Duffel Psychiatric Hospital
Locations (1):
- PZ Duffel, Duffel, Antwerp, Belgium

REFERENCES:
- [Derived] van Diermen L, Poljac E, Van der Mast R, Plasmans K, Van den Ameele S, Heijnen W, Birkenhager T, Schrijvers D, Kamperman A. Toward Targeted ECT: The Interdependence of Predictors of Treatment Response in Depression Further Explained. J Clin Psychiatry. 2020 Dec 15;82(1):20m13287. doi: 10.4088/JCP.20m13287. PMID 33326710
- [Derived] Hebbrecht K, Giltay EJ, Birkenhager TK, Sabbe B, Verwijk E, Obbels J, Roelant E, Schrijvers D, Van Diermen L. Cognitive change after electroconvulsive therapy in mood disorders measured with the Montreal Cognitive Assessment. Acta Psychiatr Scand. 2020 Nov;142(5):413-422. doi: 10.1111/acps.13231. Epub 2020 Sep 21. PMID 32895922
- [Derived] Baeten RF, Van Rossum EFC, De Rijke YB, Sabbe BGC, Van Der Mast RC, Belge JB, Fransen E, Schrijvers DL, Birkenhager TK, Van Diermen L. Hair cortisol in patients with a depressive episode treated with electroconvulsive therapy. J Affect Disord. 2020 Sep 1;274:784-791. doi: 10.1016/j.jad.2020.05.042. Epub 2020 May 28. PMID 32664015
- [Derived] Belge JB, Van Diermen L, Schrijvers D, Sabbe B, Constant E, de Timary P, De Keyzer S, Parizel P, Vansteelandt K, Sienaert P, van Eijndhoven P. The basal ganglia: A central hub for the psychomotor effects of electroconvulsive therapy. J Affect Disord. 2020 Mar 15;265:239-246. doi: 10.1016/j.jad.2020.01.033. Epub 2020 Jan 13. PMID 32090747
- [Derived] van Diermen L, Versyck P, van den Ameele S, Madani Y, Vermeulen T, Fransen E, Sabbe BGC, van der Mast RC, Birkenhager TK, Schrijvers D. Performance of the Psychotic Depression Assessment Scale as a Predictor of ECT Outcome. J ECT. 2019 Dec;35(4):238-244. doi: 10.1097/YCT.0000000000000610. PMID 31764446
- [Derived] van Diermen L, Hebbrecht K, Schrijvers D, Sabbe BCG, Fransen E, Birkenhager TK. The Maudsley Staging Method as predictor of electroconvulsive therapy effectiveness in depression. Acta Psychiatr Scand. 2018 Dec;138(6):605-614. doi: 10.1111/acps.12962. Epub 2018 Oct 1. PMID 30270433